CLINICAL TRIAL: NCT01104974
Title: Canadian Health Care Providers' Attitudes of Pregnancy, Fertility Care, and Assisted Reproductive Technologies for HIV-Positive Individuals
Brief Title: HIV Physician's Survey
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 08-310
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: HIV
Keywords: HIV; HIV providers; Infectious Disease; HIV and pregnancy
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a survey study to assess the variability in the current management of pregnancy, reproductive care and assisted reproductive technologies for HIV-positive individuals in Canada to estimate interest for further projects.

ELIGIBILITY:
Inclusion Criteria:

* any HIV health care provider

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV Providers in Canada
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)